CLINICAL TRIAL: NCT00151398
Title: A 3-Month, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Safety, Tolerability, and Efficacy Study Of 3 Doses Of Lecozotan (SRA-333) SR In Outpatients With Mild To Moderate Alzheimer's Disease With Donepezil As Active Control.
Brief Title: Study Evaluating Lecozotan SR in Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3098B1-201, 3098B1-202; B343-1057, B343-1058 (Other: Pfizer)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental)
  Interventions: Drug: lecozotan SR
- B (Experimental)
  Interventions: Drug: lecozotan SR
- C (Experimental)
  Interventions: Drug: lecozotan SR
- D (Active Comparator)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: lecozotan SR — evaluation of long term therapy with 3 doses of lecozotan sr ( 2, 5, and 10 mg)administered to patients with AD who have completed week 12 evaluations in the short-term study. Patient duration is 42 weeks.
  Arms include lecozotan sr 2 mg, 5mg, and 10 mg as well as donepezil.
  Arms: A; B; C
Drug: Donepezil — 10 mg donepezil QD dosed up to 40 weeks
  Arms: D

SUMMARY:
The purpose of this study is determine the safety, tolerability, and efficacy of 3 doses of lecozotan SR in patients with mild to moderate Alzheimer's Disease over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the NINCDS-ADRDA criteria.
* Able to give informed consent. Patient' s caregiver must consent to participate in the study.

Exclusion Criteria:

* Use of medications for cognitive enhancement within 3 months of baseline.
* Significant neurologic disease other than AD that may affect cognition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2005-10-06 (Actual); Primary Completion 2008-03-15 (Actual); Study Completion 2008-03-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoints will be the change from baseline in ADAS-Cog total score and ADCS-CGIC total score. | weeks 12, 14, 26 and 40.

SECONDARY OUTCOMES:
Secondary efficacy outcome variables include additional cognitive, functional,and behavioral measures. | weeks 12, 14, 26 and 40.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (55):
- United States (34):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Fresno, California
  - La Jolla, California
  - Orange, California
  - Boca Raton, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - St Louis, Missouri
  - Long Branch, New Jersey
  - Manchester Twp., New Jersey
  - Albany, New York
  - Cedarhurst, New York
  - Lawrence, New York
  - Staten Island, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Memphis, Tennessee
  - Houston, Texas
  - Bennington, Vermont
- Argentina (8):
  - Av. Belgrano
  - Calle Adolfo Alsina
  - Cervino
  - Gascon
  - Larrea
  - Nueva York
  - Pilar
  - Puerto Galván
- Australia (2):
  - Hornsby, New South Wales
  - Heidelberg Heights, Victoria
- Canada (6):
  - Edmonton, Alberta
  - Medicine Hat, Alberta
  - Moncton, New Brunswick
  - Ottawa, Ontario
  - Montreal, Quebec
  - Regina, Saskatchewan
- South Africa (5):
  - Westdene, Bloemfontein
  - Observatory, Cape Town
  - Panorama, Cape Town
  - Florida, Johannesburg
  - Bellville, Western Cape